CLINICAL TRIAL: NCT00554372
Title: A Phase II-a, Open-Label, Randomized Study of JX-594 (Thymidine Kinase-deleted Vaccinia Virus Plus GM-CSF) Administered by Intratumoral Injection in Patients With Unresectable Primary Hepatocellular Carcinoma
Brief Title: A Study of Recombinant Vaccinia Virus to Treat Unresectable Primary Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Organization: SillaJen, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JX594-IT-HEP007
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2011-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Jennerex; HCC; unresectable primary hepatocellular carcinoma; hepatocellular carcinoma; liver cancer; Phase 2; oncolytic virus; Pexa-Vec
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Experimental): 1e8 pfu (plaque forming units) total dose of JX-594 (recombinant vaccinia virus) on each of three (3) treatment days (2 weeks apart)
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)
- High Dose (Experimental): 1e9 pfu (plaque-forming units) total dose of JX-594 (recombinant vaccinia virus) on each of three (3) treatment days (2 weeks apart)
  Interventions: Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF)

INTERVENTIONS:
Genetic: JX-594: Recombinant vaccinia virus (TK-deletion plus GM-CSF) — Patients will be randomized 1:1 to one of two total doses (1e8 or 1e9 pfu)and injected intratumorally in 1-5 intrahepatic tumors on Days 1, 15, and 29.

SUMMARY:
The purpose of this research study is to determine whether JX-594 (Pexa-Vec) has significant anti-tumoral activity and tolerability in primary hepatocellular carcinoma and to determine the dose to be used in further testing.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is estimated to be the third most common cause of cancer-related deaths world-wide, and the fifth most common cancer diagnosis. According to the National Cancer Institute (NCI), approximately 17,000 new cases of HCC are diagnosed annually in the U.S. In Canada, the predicted incidence for 2007 is 1,350 new cases. In addition, approximately 10,000 new cases are diagnosed per year in S. Korea, 35,000 in the E.U. and 45,000 in Japan.

The five-year survival rate is estimated to be <10% for all HCC patients. Given the poor prognosis of these patients there is a desperate need for new therapies.

Surgical resection and liver transplant are the only curative treatment for HCC. Small HCC tumor(s) (less than 3 cm in diameter) can be resected by hepatectomy, the most effective treatment. Surgery was associated with a reported 50-60% five-year survival rate, but unfortunately was possible in only 10-15% of cases. Liver transplant is considered for patients with tumors that are unresectable but that are still limited exclusively to the liver, have no extracapsular or vascular invasion within the liver, and for whom there are no medical contraindications to transplantation. Patients with unresectable HCC that cannot receive liver transplantation, and who do not require systemic therapy, may be administered percutaneous ethanol injection therapy (PEIT), radiofrequency ablation (RFA), transarterial chemoembolization (TACE), and/or radioembolization, depending on the size of the intrahepatic tumors and the underlying liver function.

HCC may be a good target for IT injection with JX-594 because of the relatively high rate of accessible tumors for injection, the positive response seen in a patient with HCC in a recently completed Phase I study of JX-594 intratumoral injection within the liver, excellent tumor responses in multiple preclinical cancer models, and the lack of effective, tolerable therapy for most patients with HCC who cannot receive curative surgery or immediate liver transplantation. Furthermore, it is speculated that JX-594 replication targets the EGFR pathway, and that it's spread within and between tumors is dependent upon the intratumoral vasculature; HCC has highly activated angiogenesis and EGFR pathways in the majority of cases.

ELIGIBILITY:
Inclusion Criteria

* Histological confirmation or clinical/laboratory diagnosis of primary hepatocellular carcinoma (HCC)
* Cancer is not surgically resectable for cure
* Child Pugh A or B
* Tumor progression during or after at least one prior HCC treatment regimen (Note: If standard HCC therapies are either medically contraindicated or patient has refused those treatments, the patient may be eligible for this study)
* Performance Score: KPS score of ≥ 70
* Anticipated survival of at least 16 weeks
* Total bilirubin ≤ 2.5 x ULN
* AST, ALT < 5.0 x ULN
* WBC > 2,500 cells/mm3 and < 50,000 cells/mm3 (GCSF treatment allowed)
* ANC > 1,250 cells/mm3 (GCSF treatment allowed)
* Hemoglobin ≥ 9 g/dL (RBC transfusion allowed)
* Platelet count ≥ 50,000 plts/mm3
* Acceptable coagulation status: INR ≤ 1.5 x ULN
* Acceptable kidney function: Serum creatinine < 2.0 mg/dL
* If patients are diabetic or have a screening random glucose > 160 mg/dL, a fasting glucose must be done and patients must be WNL or Grade 1 in order to be eligible for the study
* For patients who are sexually active: able and willing to abstain from sex during treatment period and for 3 weeks following treatment, and use an acceptable method of birth control for 3 months after last injection with JX-594
* Able/willing to sign an IRB/IEC/REB-approved written consent form
* Able and willing to comply with study procedures and follow-up examinations, including compliance with the "Infection Control Guidelines for Patients" (in written consent form)

Exclusion Criteria:

* Current, known extra-hepatic tumors that, in the investigator's medical opinion, are likely to result in significant morbidity or mortality within the next 16 weeks.
* Pregnant or nursing an infant
* Known infection with HIV
* Clinically significant active infection or uncontrolled medical condition considered high risk for investigational new drug treatment
* Significant immunodeficiency due to underlying illness (e.g. hematological malignancies, congenital immunodeficiencies and/or HIV infection/AIDS) and/or medication (e.g. high-dose systemic corticosteroids)
* History of exfoliative skin condition (e.g. severe eczema, ectopic dermatitis, or similar skin disorder) that at some stage has required systemic therapy
* Clinically significant and/or rapidly accumulating ascites, peri-cardial and/or pleural effusions
* Liver tumors in a location that would potentially result in significant clinical adverse effects if post-treatment tumor swelling were to occur (e.g. tumors impinging on the biliary tract that could affect drainage)
* Severe or unstable cardiac disease
* Current, known CNS malignancy
* Anti-cancer therapy (e.g. RFA, TACE, PEIT, radioembolization, chemotherapy, surgery, or an investigational drug, etc.) within 4 weeks prior to first treatment
* Absolute contraindication to undergoing MRI scanning
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination
* Use of anti-platelet or anti-coagulation medication
* Use of the following anti-viral agents: ribavirin, adefovir, cidofovir (within 7 days prior to the first treatment), and PEG-IFN (within 14 days prior to the first treatment).
* Inability or unwillingness to give informed consent or comply with the procedures required in the protocol
* Patients with household contacts who meet any of these criteria unless alternate living arrangements can be made during the patient's active dosing period and for 7 days following the last dose of study medication:
* Pregnant or nursing an infant
* Children < 12 months old
* History of exfoliative skin condition that at some stage has required systemic therapy
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kirn, MD, Study Director — Jennerex Biotherapeutics; Tony Reid, Md, PhD, Principal Investigator — University of California San Diego, Moores Cancer Center; Jeong Heo, MD, PhD, Principal Investigator — Pusan National University
Locations (9):
- United States (5):
  - Moores UCSD Cancer Center, La Jolla, California
  - Mayo Clinic, Rochester, Minnesota
  - Billings Clinic Cancer Center, Billings, Montana
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center - Liver Cancer Center, Pittsburgh, Pennsylvania
- McMaster University Medical Centre, Hamilton, Ontario, Canada
- South Korea (3):
  - Pusan National University Hospital, Busan
  - Samsung Medical Center, Seoul
  - Shin Chon Severance Hospital / Yonsei University Medical Center, Seoul

REFERENCES:
- [Result] Heo J, Reid T, Ruo L, Breitbach CJ, Rose S, Bloomston M, Cho M, Lim HY, Chung HC, Kim CW, Burke J, Lencioni R, Hickman T, Moon A, Lee YS, Kim MK, Daneshmand M, Dubois K, Longpre L, Ngo M, Rooney C, Bell JC, Rhee BG, Patt R, Hwang TH, Kirn DH. Randomized dose-finding clinical trial of oncolytic immunotherapeutic vaccinia JX-594 in liver cancer. Nat Med. 2013 Mar;19(3):329-36. doi: 10.1038/nm.3089. Epub 2013 Feb 10. PMID 23396206
- [Derived] Breitbach CJ, Arulanandam R, De Silva N, Thorne SH, Patt R, Daneshmand M, Moon A, Ilkow C, Burke J, Hwang TH, Heo J, Cho M, Chen H, Angarita FA, Addison C, McCart JA, Bell JC, Kirn DH. Oncolytic vaccinia virus disrupts tumor-associated vasculature in humans. Cancer Res. 2013 Feb 15;73(4):1265-75. doi: 10.1158/0008-5472.CAN-12-2687. Epub 2013 Feb 7. PMID 23393196
- See also: Sponsor company website — http://www.jennerex.com
- See also: Sponsor company was acquired by SillaJen Inc. — http://www.sillajen.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized 1:1 to a treatment arm (dosage group). Randomization into the dosing groups was stratified by whether the Hepatocellular carcinoma was virally associated (hepatitis B virus or hepatitis C virus) or not virally associated.
Groups:
- Low Dose: 1e8 pfu (plaque forming units) total dose of JX-594 (recombinant vaccinia virus) on each of three (3) treatment days (2 weeks apart). Each treatment dose was divided among 1-5 hepatic tumors; all tumors injected at day 1 were also injected at subsequent treatments.
- High Dose: 1e9 pfu (plaque forming units) total dose of JX-594 (recombinant vaccinia virus) on each of three (3) treatment days (2 weeks apart). Each treatment dose was divided among 1-5 hepatic tumors; all tumors injected at day 1 were also injected at subsequent treatments.
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.5) | 62.9 (12.7) | 64.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
  Canada | 3 | 4 | 7
  Korea, Republic of | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Disease Control (Non-progressive Disease) at 8 Weeks After Initiation of Treatment
Description: Proportion of subjects achieving disease control at 8 weeks based on a modified Response Evaluation Criteria in Solid Tumors v1.0 (mRECIST). Per mRECIST for target lesions as assessed by dynamic contrast enhanced dynamic MRI: Complete Response (CR), Disappearance of all tumor(s); Partial Response (PR), >=30% decrease in the sum of longest diameter (LD) of tumor(s) taking as reference the baseline sum; Stable Disease (SD), any cases that do not qualify for PR or progressive disease (PD); PD, any increase of >= 20% in the sum of longest diameter (LD) of tumor(s) taking as reference the baseline sum. Disease Control (DC) = CR or PR or SD. For mRECIST criteria, new tumor(s) that developed within the liver were measured (a new tumor was defined as a malignant tumor not present at baseline, was ≥ 1 cm in LD had typical hypervascular features of HCC). Their maximum diameter(s) were included in the sum of the maximum diameter; new tumors were not considered evidence for progression.
Time Frame: Initial progression status and response assessment at 8 weeks from first dose
Population: Patients having evaluable radiographic imaging, 2 patients in each arm were excluded due to unevaluable images, 1 patient in the low dose arm was excluded due to a protocol deviation
Measure: Number (95% Confidence Interval); unit: Proportion of evaluable participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 13 | 15
Proportion of evaluable participants | 0.7273 [0.390 to 0.940] | 0.6429 [0.351 to 0.872]

2. Secondary Outcome: Safety and Tolerability of JX-594 Administered at Two Dose Levels
Description: Treatment-related serious adverse events in patients treated at two dose levels
Time Frame: Safety and tolerability were evaluated throughout the 8 week period of study participation
Measure: Number; unit: serious adverse event
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 14 | 16
serious adverse event | 1 | 0

3. Secondary Outcome: Number of Subjects Achieving Disease Control as Determined Using Intrahepatic Modified RECIST Criteria
Description: Number of subjects achieving disease control (non-progressive disease) at 8 weeks after treatment was initiated based on modified Response Evaluation Criteria in Solid Tumors for Hepatocellular Carcinoma (mRECIST for HCC). mRECIST for HCC adopted the concept of viable tumor as tumor tissue showing uptake in arterial phase of contrast enhanced radiologic imaging techniques. (see Lencioni and Llovet, Semin. Liver Dis. 2010; 30:52-60). Per mRECIST for HCC, for target lesions as assessed by contrast enhanced dynamic MRI: Complete Response (CR), Disappearance of any intratumoral arterial enhancement in all target (viable) lesions; Partial Response (PR), >=30% decrease in the sum of diameters of viable target lesions; Stable Disease (SD), any cases that do not qualify for PR or progressive disease (PD); PD, any increase of >= 20% in viable target lesions.
  Disease Control (DC) = CR or PR or SD.
Time Frame: At week 8
Measure: Number; unit: participants
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 13 | 15
participants | 6 | 7

4. Secondary Outcome: Median Overall Survival
Description: Overall survival after treatment in days
Time Frame: To 760 days post treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 13 | 16
days | 202 [109 to 271] | 423 [265 to NA] — Upper bound was not achieved. The data analysis was done at a time when subjects in both dose groups were still alive.

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 4/14 | 4/16
Other Adverse Events (participants affected / at risk) | 14/14 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=14) | High Dose (N=16)
Bile duct Obstruction (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 (0)
Angina pectoris (Cardiac disorders) | 1 | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1
Vomiting (Gastrointestinal disorders) | 0 (0) | 1
Bacteraemia (Infections and infestations) | 1 | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=14) | High Dose (N=16)
Lymphopenia (Blood and lymphatic system disorders) | 4 | 3
Tachycardia (Cardiac disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 5 | 8
Vomiting (Gastrointestinal disorders) | 8 | 6
Abdominal Pain (Gastrointestinal disorders) | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Pyrexia (General disorders) | 13 | 16
Chills (General disorders) | 11 | 13
Influenza like illness (General disorders) | 4 | 4
Injection site pain (Injury, poisoning and procedural complications) | 6 | 9
Fatigue (General disorders) | 4 | 6
Asthenia (General disorders) | 1 | 2
Hyperbilirubinemia (Hepatobiliary disorders) | 2 | 2
Hemoglobin Decreased (Investigations) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 5 | 6
Confusional state (Psychiatric disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Edema peripheral (General disorders) | 3 | 1
Chest Discomfort (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 5
Abdominal Pain (lower) (Gastrointestinal disorders) | 2 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 1
Stomach Discomfort (Gastrointestinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferse increased (Investigations) | 4 | 1
Lymphocyte count decreased (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood Alkaline Phosphatase increased (Investigations) | 1 | 1
Hemoglobin (Investigations) | 1 | 2
Hematocrit decreased (Investigations) | 1 | 1
Platelet Count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 4
Muscoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days